CLINICAL TRIAL: NCT05199779
Title: A Single Session Intervention Leveraging an Ultra-Brief Exercise for Building Self-Compassion Habits-A Randomized Controlled Trial
Brief Title: Single Session Intervention for Building Self-Compassion Habits-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Responsible Party: Principal Investigator, Allison Harvey, Professor of Clinical Psychology, University of California, Berkeley
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-12-14924
Record Dates: First submitted 2022-01-05; First posted 2022-01-20 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Transdiagnostic Psychopathology
Keywords: Self-Compassion; Habits; Transdiagnostic; Intervention
MeSH Terms: conditions — Habits

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to the SCI or AC control using the randomizer elements in Qualtrics.
Who Masked: Participant
Masking Description: To reduce bias in the assessments, none of the constructs of interest to this study (e.g., "stress", "self-compassion") will be included in the language used to describe the intervention or in any materials used to advertise the study. Study participants will be told they are participating in a study on "fostering emotional well-being". No further information about the intervention will be provided.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-Compassion Intervention (SCI) (Experimental): First, participants will be taught to implement a 20-second self-compassion induction via video recording. Second, participants will be taught to choose a cue that will precede their daily use of the self-compassion induction. Participants will document the cue they chose, and will be emailed a record of their selected cue, along with the recording and transcript of the self-compassion induction that they can refer back to for reference. Third, participants will be asked to use the self-compassion induction as much as they can and at least once during their daily routine following exposure to their chosen cue.
  Interventions: Behavioral: Single Session Intervention Leveraging an Ultra-Brief Self-Compassion Exercise
- Finger-Tapping Active Control (AC) (Active Comparator): The active control will receive the same procedures as described above, except for receiving a different video containing different instructions describing a finger-tapping exercise. The videos will be virtually identical in length, quality, instructor/their outfit, and lighting.
  Interventions: Behavioral: Finger-Tapping Active Control

INTERVENTIONS:
Behavioral: Single Session Intervention Leveraging an Ultra-Brief Self-Compassion Exercise — This 20-second contemplative exercise includes draws from the science of habit formation and includes elements of self-soothing touch, somatic experiencing, and mindful self-compassion.
  Arms: Self-Compassion Intervention (SCI)
Behavioral: Finger-Tapping Active Control — This 20-second finger tapping exercise involves touching each finger to the thumb on one hand and repeating for twenty seconds. This intervention was designed to control for the potential effect of assessment on outcomes, the effect of having an activity to do for the duration of the intervention (4 weeks), regression to the mean, time, or other nonspecific factors.
  Arms: Finger-Tapping Active Control (AC)

SUMMARY:
The study will test a single session self-compassion intervention that leverages an ultra-brief contemplative exercise. It will evaluate the effect of this intervention on psychopathology, stress, growth mindset, positive affect, self-compassion and the automaticity of self-compassion, as well as the relationships between these constructs and the automaticity of self-compassion. The participants will be undergraduate students at a large public university.

DETAILED DESCRIPTION:
The broad aims of the proposed research is to examine the outcomes of a single session psychological intervention and to further understand processes and factors associated with habit formation. undergraduate students at a large university will be randomly assigned to a self-compassion intervention (SCI), or an active control (AC), and complete assessments at baseline (pre-treatment) and 4 weeks later (post-treatment).

The investigators seek to examine the following: (A1) Determine whether the group who receives the SCI, relative to the AC, will experience increased self-compassion, growth mindset and positive affect, as well as reduced stress and psychopathology. (A2) Evaluate whether the SCI group shows greater increases in automaticity of self-compassion compared to the AC pre- to post-treatment. (A3) Assess whether greater pre- to post-treatment increases in automaticity of self-compassionate are associated with increased self-compassion, growth mindset, and positive affect, as well as reductions in stress and psychopathology.

The investigators hypothesize the following: (H1) SCI will promote greater increases in self-compassion, growth mindset, and positive affect, as well as greater reductions in stress and psychopathology from pre- to post-treatment, relative to AC. (H2) The SCI group will show greater increases in the automaticity of self-compassion than AC from pre- to post-treatment. (H3) Greater increases in the automaticity of self-compassion from pre- to post-treatment will be predicted by greater increases in self-compassion, growth mindset, and positive affect, as well as greater decreases in psychopathology and stress, from pre- to post treatment. To further understand the results obtained, the investigators will evaluate participants' frequency, adherence, and impressions of using the intervention.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* English language proficiency.
* Able and willing to give informed consent.

Exclusion Criteria:

* Does not have email address or access to email.
* Not able/willing to participate in and/or complete the pre-treatment assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2022-02-13 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
Sussex-Oxford Compassion for the Self Scale (SOCS-S) | Change from baseline to post-treatment (week 4)
  Sum of 20-item, 5-point response scale. Scores can range from 20 to 100 (Higher score means higher compassion for self).
  Sub-scale items included.
Kind of Person' Implicit Theory Scale (KOPITS) | Change from baseline to post-treatment (week 4)
  8 items. 6-point response scale (1 = strongly agree; 6 = strongly disagree) Higher scores indicate a more growth mindset. Lower scores indicate a more fixed mindset.
  Score is sum of all items, with Q3, Q5, Q7, and Q8 reverse-scored. The formula for reverse-scoring an item is: ((Number of scale points) + 1) - (Respondent's answer)
Positive and Negative Affect Schedule (PANAS) | Change from baseline to post-treatment (week 4)
  10 items with a 6 point response scale. Positive affect sub-scale only.
  Scoring:
  Positive Affect Score: Sum score of 1, 3, 5, 9, 10, 12, 14, 16, 17, and 19. Scores range from 10 - 50. Higher scores = higher levels of positive affect.
  Negative Affect Score: Sum score of 2, 4, 6, 7, 8, 11, 13, 15, 18, and 20. Scores range from 10 - 50. Lower scores = lower levels of negative affect.
10-item Perceived-Stress Scale (PSS-10) | Change from baseline to post-treatment (week 4)
  10 items, 5 point response scale (from 0 = Never to 4 = Very Often)
  Scoring: Reverse score (e.g., 0 = 4, 1 = 3, 2 = 2, 3 = 1 & 4 = 0) items 4, 5, 7, & 8 and then summing across all scale items.
DSM-5 Cross-Cutting Measure (DSM-XC) | Change from baseline to post-treatment (week 4)
  22 items (suicidality item Q11 removed). 5-point scale (0=none or not at all; 1=slight or rare, less than a day or two; 2=mild or several days; 3=moderate or more than half the days; and 4=severe or nearly every day).
Self-Report Behavioral Automaticity Index for Self-Compassion | Change from baseline to post-treatment (week 4)
  20 items. 1-9 scale.

SECONDARY OUTCOMES:
State Self-Compassion Scale Long Form (SSCS-L) | Change from pre-induction to post-induction at baseline and at post-treatment (week 4). Change in pre to post-induction changes in state self-compassion from baseline to post-treatment (week 4)
  9 items. 1-5 scale. Scores range from 9-45. Mindfulness, common humanity, and self-kindness sub-scales only.
Self-Report Behavioral Automaticity Index for Exercise | Change from baseline to post-treatment (week 4)
  4 items. 1-9 scale.
Real Self Overlap Scale | Change from baseline to post-treatment (week 4)
  1 item. 1-8 scale.

OTHER OUTCOMES:
Practice Frequency | Assessed at Post-treatment (week 4)
  Number of times practiced self-compassion exercise per day. 1 item.
Overall Practice Frequency | Assessed at Post-treatment (week 4)
  Number of days in the past two months that did not practice the exercise at all. 1 item.
Practice Duration | Assessed at Post-treatment (week 4)
  1 item, number of days practiced exercise but for less than 10 seconds.
Adherence Report Scale | Assessed at Post-treatment (week 4)
  10 items on a five-point scale, where 5 = never, 4 = rarely, 3 = sometimes, 2 = often and 1 = always. Scores for each item were summed to give a total score, with higher scores indicating higher levels of reported adherence.
General impressions of exercise | Assessed at Post-treatment (week 4)
  Exploratory qualitative assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Allison Harvey, PhD, Principal Investigator — University of California, Berkeley; Eli S Susman, BA, Principal Investigator — University of California, Berkeley
Locations (1):
- University of California at Berkeley, Berkeley, California, United States

REFERENCES:
- [Derived] Susman ES, Chen S, Kring AM, Harvey AG. Daily micropractice can augment single-session interventions: A randomized controlled trial of self-compassionate touch and examining their associations with habit formation in US college students. Behav Res Ther. 2024 Apr;175:104498. doi: 10.1016/j.brat.2024.104498. Epub 2024 Feb 21. PMID 38412573